CLINICAL TRIAL: NCT00004901
Title: A Phase I Study of Concomitant Chemoradiotherapy With 776C85, 5-FU and Hydroxyurea for Patients With Poor Prognosis Oral Cancer
Brief Title: Combination Chemotherapy Plus Radiation Therapy in Treating Patients With Advanced Mouth Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Robert H. Lurie Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: NU-V95N4; CDR0000067580 (Registry Identifier: PDQ (Physician Data Query)); NCI-G00-1680
Record Dates: First submitted 2000-03-07; First posted 2004-07-26 (Estimated); Last update posted 2013-06-26 (Estimated); Status verified 2000-08

CONDITIONS: Head and Neck Cancer
Keywords: stage IV hypopharyngeal cancer; recurrent hypopharyngeal cancer; stage IV squamous cell carcinoma of the lip and oral cavity; stage IV verrucous carcinoma of the oral cavity; stage IV mucoepidermoid carcinoma of the oral cavity; stage IV adenoid cystic carcinoma of the oral cavity; recurrent squamous cell carcinoma of the lip and oral cavity; recurrent verrucous carcinoma of the oral cavity; recurrent mucoepidermoid carcinoma of the oral cavity; recurrent adenoid cystic carcinoma of the oral cavity; stage IV squamous cell carcinoma of the oropharynx; stage IV lymphoepithelioma of the oropharynx; recurrent squamous cell carcinoma of the oropharynx; recurrent lymphoepithelioma of the oropharynx; stage IV squamous cell carcinoma of the nasopharynx; stage IV lymphoepithelioma of the nasopharynx; recurrent squamous cell carcinoma of the nasopharynx; recurrent lymphoepithelioma of the nasopharynx; stage IV squamous cell carcinoma of the hypopharynx; recurrent squamous cell carcinoma of the hypopharynx; stage IV squamous cell carcinoma of the larynx; stage IV verrucous carcinoma of the larynx; recurrent squamous cell carcinoma of the larynx; recurrent verrucous carcinoma of the larynx
MeSH Terms: conditions — Head and Neck Neoplasms; Hypopharyngeal Neoplasms; Squamous Cell Carcinoma of Head and Neck | interventions — eniluracil; Fluorouracil; Hydroxyurea; Radiotherapy

INTERVENTIONS:
Drug: ethynyluracil
Drug: fluorouracil
Drug: hydroxyurea
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Radiation therapy uses high-energy x-rays to damage tumor cells. Combining more than one chemotherapy drug with radiation therapy may kill more tumor cells.

PURPOSE: Phase I/II trial to study the effectiveness of combination chemotherapy plus radiation therapy in treating patients who have advanced mouth cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Assess the feasibility of the administration of ethynyluracil concurrently with fluorouracil and radiotherapy in patients with advanced oral cancer. II. Determine the maximum tolerated dose (MTD) and dose-limiting toxicities of this regimen in this patient population.

OUTLINE: This is a dose escalation study of fluorouracil and hydroxyurea. Patients receive oral ethynyluracil every 12 hours on days 1-7 and oral fluorouracil every 12 hours on days 2-6. Radiotherapy to the head and neck is administered twice daily on days 2-6. Treatment continues for 5-7 courses in the absence of unacceptable toxicity. Cohorts of 3-6 patients receive escalating doses of fluorouracil until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 3 of 6 patients experience dose limiting toxicities. Once the MTD of fluorouracil is determined, hydroxyurea is added to the treatment regimen. Patients receive fluorouracil and ethynyluracil as per the treatment schedule outlined above. Patients also receive oral hydroxyurea every 12 hours for 11 doses on days 1-6. Radiotherapy is administered as above. Cohorts of 3-6 patients receive escalating doses of hydroxyurea until the MTD is determined. Once the MTD of fluorouracil and hydroxyurea are determined, an additional 10 patients receive Phase II doses of ethynyluracil, fluorouracil and hydroxyurea as per the treatment schedule outlined above. Treatment continues in the absence of unacceptable toxicity. Patients are followed at 4-6 weeks, then every 6 months until death.

PROJECTED ACCRUAL: Approximately 40 patients will be accrued for this study over 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically or cytologically confirmed advanced malignant oral or laryngeal neoplasm requiring regional radiotherapy and not amenable to standard therapy Tumor site amenable to radiotherapy

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: ECOG 0-2 Life expectancy: Expected 2 year survival less than 10% in previously untreated patients Hematopoietic: WBC at least 3,000/mm3 Platelet count at least 100,000/mm3 Hepatic: Not specified Renal: Creatinine clearance at least 50 mL/min Other: No severe infection or medical illness that would preclude study Must be able to swallow and retain oral medications Not pregnant

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: Recovered from prior chemotherapy Endocrine therapy: Not specified Radiotherapy: Recovered from prior radiotherapy Surgery: Not specified

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1999-10; Study Completion 2004-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Everett E. Vokes, MD, Study Chair — University of Chicago
Locations (2):
- United States (2):
  - Robert H. Lurie Comprehensive Cancer Center, Northwestern University, Chicago, Illinois
  - University of Chicago Cancer Research Center, Chicago, Illinois